CLINICAL TRIAL: NCT05129111
Title: A Stimulator of the Salivary Excretion Based on Physical Vibration of the Parotid Glands.
Brief Title: A Stimulator of the Salivary Vibration of the Parotid Glands
Acronym: saliva
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Pia Lopez Jornet, Investigador principal, Universidad de Murcia
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3338/2021
Record Dates: First submitted 2021-11-01; First posted 2021-11-22 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Saliva Stimulated
Keywords: saliva

STUDY DESIGN:
Intervention Model Description: The central idea of the device resides in transmitting the vibration generated by two vibrating modules to the two parotid glands through the superficial contact established between each vibrating module and the respective parotid gland, achieving the stimulation of both parotid glands simultaneously.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- STIMULATOR OF THE SALIVARY EXCRETION BASED ON PHYSICAL VIBRATION (Active Comparator): Measurement of salivary secretion at rest and stimulated conditions.
  Interventions: Device: PHYSICAL VIBRATION OF THE PAROTID GLANDS
- STIMULATOR OF THE SALIVARY EXCRETION PLACEBO (Placebo Comparator): Measurement of salivary secretion at rest and stimulated conditions.
  Interventions: Device: PHYSICAL VIBRATION OF THE PAROTID GLANDS

INTERVENTIONS:
Device: PHYSICAL VIBRATION OF THE PAROTID GLANDS — The system will be placed bilaterally in the parotid glands and assessed the efficacy of the salivary secretion by sialometry before and after the stimulation

SUMMARY:
Oral dryness causes significant health problems both functional (difficulty speaking, chewing and swallowing) and structural problems in teeth (increased number of infections) and oral mucosa. The main objective of this study is to show an alternative treatment to help to stimulate the salivary secretion thus improving the quality of life of the patient. In this study, a salivary stimulation equipment using vibrotactile stimuli is shown. The system has been placed bilaterally in the parotid glands and assessed the efficacy of the salivary secretion by sialometry before and after the stimulation. The new proposal is capable of stimulating salivary secretion, in a significative way after 7 minutes of use, at least in the cases analyzed, and fulfills low-cost, easy-to-use and safe technical restrictions. In this setting, this paper suggests the performance of a deep clinical trial to measure the exact efficacy of the prototype and the times and frequencies needed to state the optimal treatment depending in each case

ELIGIBILITY:
Inclusion Criteria:

* Sialometria <01,mL /5 min
* Test Thomson

Exclusion Criteria:

* Not signing informed consent
* Bad medical status

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2021-07-03 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
sialometry | up to 4 weeks
  The test we will use consists of measuring the amount of saliva produced during a period of 5 mins when a millimetre strip of paper with a dimension of 1 cm wide and 17 cm is applied.

CONTACTS AND LOCATIONS:
Locations (1):
- Lopez-Jornet Pia, Murcia, N/A = Not Applicable, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fernandes MS, Castelo PM, Chaves GN, Fernandes JPS, Fonseca FLA, Zanato LE, Gaviao MBD. Relationship between polypharmacy, xerostomia, gustatory sensitivity, and swallowing complaints in the elderly: A multidisciplinary approach. J Texture Stud. 2021 Apr;52(2):187-196. doi: 10.1111/jtxs.12573. Epub 2020 Nov 25. PMID 33191538
- [Background] Salimi F, Saavedra F, Andrews B, FitzGerald J, Winter SC. Trans-cutaneous electrical nerve stimulation to treat dry mouth (xerostomia) following radiotherapy for head and neck cancer. A systematic review. Ann Med Surg (Lond). 2021 Feb 3;63:102146. doi: 10.1016/j.amsu.2021.01.094. eCollection 2021 Mar. PMID 33664943